CLINICAL TRIAL: NCT04582331
Title: Improving Real-time COVID-19 Monitoring Through Smartphone Voice Analysis
Status: Completed | Type: Observational
Sponsor: Sonde Health (Industry)
Responsible Party: Sponsor
Other Study IDs: SH2020.COV01
Record Dates: First submitted 2020-10-07; First posted 2020-10-09 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Covid19
Keywords: Respiratory disease; Respiratory infection; Vocal biomarkers; Digital health; Symptom monitoring
MeSH Terms: conditions — COVID-19; Respiration Disorders; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID-19 positive: Patients with suspected COVID-19 based on presence of at least one newly emerged relevant symptom that has emerged at most 10 days prior to enrollment. COVID-19 positive status is confirmed by diagnostic testing and clinical diagnosis.
  Interventions: Other: Smartphone-based voice and self-reported symptom collection
- COVID-19 negative, symptomatic: Patients with suspected COVID-19 based on presence of at least one newly emerged relevant symptom that has emerged at most 10 days prior to enrollment. COVID-19 negative status is confirmed by diagnostic testing and clinical diagnosis.
  Interventions: Other: Smartphone-based voice and self-reported symptom collection
- Normal Healthy Volunteers: Asymptomatic healthy participants recruited from hospital staff or co-living family members, or co-living family member of a COVID-19 positive study participant.
  Interventions: Other: Smartphone-based voice and self-reported symptom collection

INTERVENTIONS:
Other: Smartphone-based voice and self-reported symptom collection — Voice samples and COVID-19 symptom inventories will be collected on participant smartphone devices. No outcomes or feedback is provided on acquired data during trial conduct but will be used for confirmatory data analysis post study

SUMMARY:
This is a confirmatory study that seeks to examine whether respiratory-responsive vocal biomarkers have potential to respond to COVID-19 infection status and respiratory symptom severity. Patients with suspected COVID-19 and healthy controls will submit daily voice samples and symptom inventories on their personal smartphone devices for 14 days.

DETAILED DESCRIPTION:
This is an observational study examining the potential to use voice analysis to aid in the identification of COVID-19 and as an aid to monitoring of respiratory symptoms of COVID-19. Patients with suspected COVID-19 and healthy controls will be enrolled and use their own smartphone device to provide daily voice samples and symptom inventories. This study seeks to confirm and extend findings from preliminary data from patients with asthma, COPD and cough that has indicated the potential of respiratory responsive vocal biomarkers (RRVB) to respond to respiratory diagnoses and symptom severity. The same RRVB will be examined to confirm whether this potential generalizes to respiratory symptoms associated with COVID-19

ELIGIBILITY:
Inclusion Criteria:

1. Own an eligible smartphone (iOS or Android) that is able to download and run the Sonde Health app (access to smartphone provided by parent or legal guardian of participants under the age 18 is allowed)
2. Willing to sign up for a Sonde app account
3. Agreement with the subject consent information presented on the Sonde app. In case of adolescent subjects, agreement with subject consent information provided by a parent or legal guardian
4. Stated willingness and ability to comply with all study procedures for the duration of the study
5. Male or female, aged 12 or above (including adults)
6. Able to read and speak English or Spanish (required to follow app instructions and provide correct voice elicitations)
7. Pregnant women are allowed to participate

   For suspected COVID-19 patients:
8. Confirmed or suspected COVID-19 infection with mild or severe illness severity at screening on Day 1
9. Suspected COVID-19 includes patients having at least one of the following symptoms that are present at most 10 days prior to enrollment:

   * Cough
   * Fever (>37.5 C/ 99.5 F)
   * Shortness of breath
   * Sore throat
   * Diarrhea
   * Anosmia
   * Loss of taste/ ageusia
10. COVID-19 viral test ordered at the study site within at most 5 days prior to or on Day 1

    For healthy volunteers:
11. Hospital staff or co-living family members, or co-living family member of a COVID-19 positive patient that is enrolled in this study
12. Age 12 and above

Exclusion Criteria:

1. Difficulties with speech production
2. Difficulties reading or responding to instructions and questions on a smartphone screen
3. Critical COVID-19 illness severity at screening on Day 1
4. Other critical health condition where study participation would place unreasonable burden or risk on the patient as determined by the study site principal investigator

   For healthy volunteers:
5. History of positive COVID-19 viral or serologic test result any time prior to enrollment
6. Any hospital staff that is a member of the study team, and staff in the pulmonary and infectious disease departments of the participating institution, or any of their co-living family members

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting with suspected COVID-19 with mild or severe disease severity.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
Vocal biomarker performance in COVID-19 positive vs. healthy controls | Day 1 of study enrollment
  Sensitivity, Specificity and Diagnostic Odds Ratio of RRVB, either alone or in combination with a symptom inventory, to identify COVID-19 positive patients vs. asymptomatic healthy controls

SECONDARY OUTCOMES:
Vocal biomarker vs. symptom burden correlation in COVID-19 positive | Pooled across study Days 1-14
  Mean and 90% confidence interval of the correlation coefficient distribution between RRVB-based scores and self-reported respiratory symptom burden pooled across study days within individual COVID-19 patients
Vocal biomarker performance in COVID-19 positive vs. COVID-19 negative symptomatic | Day 1 of enrollment
  Sensitivity, Specificity and Diagnostic Odds Ratio of RRVB, either alone or in combination with a symptom inventory, to discriminate COVID-19 positive vs. symptomatic COVID-19 negative patients on Day 1

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - UC San Diego Medical Center, San Diego, California
  - Brigham & Woman's Hospital, Boston, Massachusetts
  - Montefiore Medical Center, New York, New York
- Deenanath Mangeshkar Hospital & Research Centre, Pune, India

IPD SHARING:
Plan to Share IPD: No